CLINICAL TRIAL: NCT05668234
Title: Study of the Parent's Subjective Experience Following a Parent-child Psychotherapy by Interactive Guidance or Integrative Psychodynamic Psychotherapy.
Brief Title: Study of the Parent's Subjective Experience of Parent-child Psychotherapy.
Acronym: ESPPRI
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/731
Record Dates: First submitted 2022-12-09; First posted 2022-12-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Subjective Experience of Parent-child Psychotherapy
Keywords: parent-child psychotherapy; semi-structured interview
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents: Parent having carried out and completed parent-child psychotherapy with a child in CHU Minjoz (child under 5 years old).
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — semi-directive interview

SUMMARY:
The child psychiatric care of children under age of 5 years involves taking care of the child, the parent and their interaction. The investigators know that the parent-child relationship plays a key role in attachment and the mental and cerebral development of the child and many studies have shown that the interaction based psychotherapy allows an improvement in the symptoms of the child. The aim of this qualitative and exploratory study is to evaluate the parent's subjective experience of the parent-child psychotherapeutic treatment, i.e., evaluate their experience of the psychotherapy, their relationship with the therapist and a possible change occurring during the psychotherapy. The analysis will be based on semi-structured interviews that will be carried out with the parents.

DETAILED DESCRIPTION:
Parent-child psychotherapy is the first-line treatment in the context of a dysfunctional parent-child interaction and takes into account both the parent's skills/fragilities, the child's modes of expression of suffering, and their relational modalities.

The care of the parent-child interaction has been the subject of many studies, but has rarely been evaluated from the point of view of the parent, even if the latter is one of the main actors in this interaction.

In France, about 50% of the parent-child psychotherapeutic treatments lead to clinical improvement. They are mainly based on the use of integrative psychodynamic psychotherapies (PPI). PPIs, based on speech, allow the therapist to identify conflicts or anxieties related to the past or present history of the parents and to relate the current troubles of the child to these conflicts of the past. This requires sufficiently significant capacities of narration and mentalization (which consists in the capacity to intellectualize one's own psychic conflicts). The literature shows that for 50% of the population, this treatment does not seem to allow engagement in care. It is important to also explore the relationship between therapist and subject, central element in psychotherapies, and the notion of therapeutic alliance from the subject's point of view. This study aims to evaluate the subjective experience of the parents, following parent-child psychotherapy. The investigaotors consider that the parents are experts in their experience and that the interviews can help them better understand the therapeutic process of the parent-child psychotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Parent having carried out and completed parent-child psychotherapy with a child in the CHU Minjoz (child under 5 years old)
* Fluent in French.
* Not having expressed his opposition to participate.
* Affiliation to a French social security scheme or beneficiary of such affiliation.

Exclusion Criteria:

* Parent suffering from a severe and untreated psychiatric illness.
* Parent and/or dyad benefiting from psychiatric care in a day hospital and/or in full hospitalization
* Parent whose child has autism or neurodevelopmental disorders.
* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Subject without health insurance
* Pregnant woman
* Subject being in the period of exclusion from another study or declared in the "national volunteer file".

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parents who have benefited from psychotherapy treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
perception of change | 6 months
  Evaluate perception of change using a semi-structured interviews
Different ability to mentalize and understand the difficulties that had led to a request for psychotherapy | 6 months
  Evaluate ability to mentalize and understand the difficulties that had led to a request for psychotherapy using a semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Monika Szymanska, PhD, Study Chair — Centre Hospitalier Universitaire de Besancon; Livia Vicentini, Study Chair — Centre Hospitalier Universitaire de Besancon; Aline Chassagne, PhD, Study Chair — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU de besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No